CLINICAL TRIAL: NCT04165993
Title: Phase II Study of Efficacy and Safety Evaluation of KN026 Monotherapy or Combination Therapy in Patients With HER2 Expressing or Positive Metastatic Breast Cancer
Brief Title: Study of KN026 Monotherapy or Combination Therapy in Patients With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KN026-201
Record Dates: First submitted 2019-11-01; First posted 2019-11-18 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Concurrent chemotherapy and KN026 (Experimental): KN026 combined with docetaxol
  Interventions: Drug: Concurrent chemotherapy and KN026
- KN026 monotherapy (Experimental): KN026 monotherapy
  Interventions: Drug: KN026 monotherapy
- A combination treatment of KN026 and KN046 (Experimental): KN026 combined with KN046
  Interventions: Drug: KN026 combination

INTERVENTIONS:
Drug: Concurrent chemotherapy and KN026 — 30 mg/kg Q3W KN026 75 mg/m2 docetaxol
  Other Names: docetaxol
  Arms: Concurrent chemotherapy and KN026
Drug: KN026 monotherapy — 30 mg/kg Q3W KN026
  Other Names: KN026
  Arms: KN026 monotherapy
Drug: KN026 combination — 30 mg/kg Q3W KN026 5 mg/kg Q3W KN046
  Other Names: KN046
  Arms: A combination treatment of KN026 and KN046

SUMMARY:
This is an open-label, three-cohort phase 2 study of KN026 in subjects with advanced breast Cancer.

DETAILED DESCRIPTION:
KN026 is an anti-HER2 bispecific antibody that can simultaneously bind two non-overlapping epitopes of HER2, leading to a dual HER2 signal blockade.The HER2- positive mBC subjects without systemic treatment will be enrolled in cohort 1 and received 30 mg/kg KN026 and docetaxol. The HER2 low expression and hormone-receptor positive mBC subjects failed standard chemotherapy and hormone therapy will be enrolled in cohort 2 and received 30 mg/kg KN026 monotherapy. The HER2 low expression and hormone-receptor negative/weak positive mBC subjects failed standard chemotherapy will be enrolled in cohort 3 and received 30 mg/kg KN026 and 5 mg/kg KN046

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject >= 18 years
* Histologically/cytologically confirmed, locally advanced unresectable or metastatic breast cancer
* ECOG score 0 or 1
* Life expectancy >3 months
* According to the definition of RECIST1.1, the patient has at least one measurable lesion
* Adequate organ function prior to start treatment with KN026
* Able to understand, voluntarily participate and willing to sign the ICF

Exclusion Criteria:

* Accepted any other anti-tumor drug therapies within 4 weeks before fist dose
* Accepted radiotherapy within 4 weeks before enrollment
* Subjects are eligible with clinically controlled and stable neurologic function >= 4 weeks, which is no evidence of CNS disease progression; Subjects with spinal cord compression and cancerous meningitis are not eligible
* Pregnant or nursing females；or intend pregnancy within this study period or within 6 monthes after the end of this study
* History of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation
* History of immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or a history of organ transplantation
* Cavity effusion (pleural effusion, ascites, pericardial effusion, etc.) are not well controlled, and need locally treatment or repeated drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Throughout the duration of the study; up to 2 years
  Objective response rate (ORR) per RECIST 1.1 criteria according to investigators assessment
Duration of response (DOR) | up to 2 years
  Duration of response (DOR) per RECIST 1.1 criteria according to investigators assessment

SECONDARY OUTCOMES:
Percentage of participants with adverse events (AEs), serious adverse events (SAEs) and AEs of special interest | Throughout the duration of the study
  AEs, SAEs
Progression free survival (PFS) rates | 6 months and 12 months
  Progression free survival (PFS) rates
Overall survival (OS) rates | 6 months and 12 months
  Overall survival (OS) rates
durable benefit rate (DBR) | DBR calculated as the proportion of subjects with best overall response of CR, PR, or SD ≥24 weeks
  durable benefit rate (DBR)

CONTACTS AND LOCATIONS:
Overall Officials: Qingyuan Zhang, Professor, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No